CLINICAL TRIAL: NCT01163461
Title: Real Word Effects in Phonological Treatment for Word Retrieval
Brief Title: Phonomotor Treatment of Word Retrieval Deficits in Individuals With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C6572-R
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment (Experimental): individuals will receive 60 hours of speech therapy
  Interventions: Behavioral: speech therapy
- Delayed Treatment (Experimental): individuals will receive 60 hours of speech therapy after 6 week delay period
  Interventions: Behavioral: speech therapy

INTERVENTIONS:
Behavioral: speech therapy — individuals will receive 60 hours of behavioral speech therapy

SUMMARY:
This is a behavioral speech therapy trial for individuals who have suffered a stroke on the left side of the brain and have difficulty speaking. The name of this disorder is called 'aphasia'. Individuals who participate in this study will receive 60 hours of therapy for free (2 hours/day, 5 days/week, 6 weeks).

DETAILED DESCRIPTION:
The study design was a single group (n=26) with repeated testing (3 times) pre- and post-treatment. All participants received the same treatment protocol (described in detail in Appendix A and in Minkina et al. (under review)). In order to control for improvement in language function related to passage of time, and for the effect of repeated exposure to outcome measures, individuals were randomly assigned to one of two conditions: delayed treatment or immediate treatment (Figure 2). Participants who were randomized to the delayed group received repeated testing three times before and three times after a six-week delay. During the delay phase they were permitted to participate in usual speech-language care (e.g., conversation groups and individual therapy).

Standardized assessments and outcome measures (described in detail below) were administered prior to the start of treatment (for both immediate and delayed groups), at the end of the delay phase (delayed group only), immediately after treatment termination, and at three months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* left hemisphere stroke
* monolingual English speaking
* right handed
* presence of aphasia

Exclusion Criteria:

* preexisting neurological condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2014-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. Kendall, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendall DL, Hunting Pompon R, Brookshire CE, Minkina I, Bislick L. An analysis of aphasic naming errors as an indicator of improved linguistic processing following phonomotor treatment. Am J Speech Lang Pathol. 2013 May;22(2):S240-9. doi: 10.1044/1058-0360(2012/12-0078). PMID 23695900

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed Aphasia Therapy: 14 individuals were randomized to received aphasia therapy following a 6-week control delay phase. Upon completion of the 6-week control phase, they received 60 hours of behavioral therapy
- Immediate Aphasia Therapy: 14 individuals were randomized to received 60 hours of aphasia therapy immediately following testing. (no delay)
Period: Overall Study
Arm/Group | Delayed Aphasia Therapy | Immediate Aphasia Therapy
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Aphasia Therapy: Single group, open trail where 28 individuals with aphasia received 60 hours of therapy
Arm/Group | Behavioral Aphasia Therapy
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Speech Production
Description: percent change in the number of untrained words spoken correctly
Time Frame: Baseline to one week post treatment termination and three months post treatment termination
Measure: Mean (Standard Deviation); unit: % change score of untrained real words
Arm/Group | Behavioral Aphasia Therapy
Number analyzed (Participants) | 28
% change score of untrained real words
  % change immediately post treatment | 5.27 (8.09)
  % change 3 months post treatment | 5.28 (7.55)

ADVERSE EVENTS:
Groups:
- Single Group Open Trial: 28 individuals were randomized to receive either immediate speech therapy, or delayed speech therapy (following a 6 week delay period to control for Hawthorne effects). All participants received 60 hours of speech therapy 2 hours/day, 5 days/week for 6 weeks. Language behaviors were testing before, after and 3 months later.
Arm/Group | Single Group Open Trial
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Group Open Trial (N=28)
No adverse events (Social circumstances) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes